CLINICAL TRIAL: NCT02327676
Title: Emtricitabine for Naive Child Chinese Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asian-Pacific Alliance of Liver Disease, Beijing (Other)
Collaborators: Beijing Ditan Hospital (Other); Hebei Medical University Pharmaceutical Factory (Industry); National Health and Family Planning Commission, P.R.China (Other Government)
Responsible Party: Principal Investigator, Jun Cheng, chaireman of Asian-Pacific Alliance of Liver Diseas,Beijing, Asian-Pacific Alliance of Liver Disease, Beijing
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FTC-01-child patients
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Hepatitis B, Chronic
Keywords: Hepatitis B, chronic; Emtricitabine; Child
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- naive child CHB group (Experimental): 200 patients take generic emtricitabine capsule(200 mg one time per day) for 48 weeks
  Interventions: Drug: Emtricitabine

INTERVENTIONS:
Drug: Emtricitabine — emtricitabine were given to each patients for 48 weeks
  Other Names: Brand name：Huierding

SUMMARY:
This study evaluates generic emtricitabine(FTC) in Chinese naive children chronic hepatitis B patients. Single group of child patients were enrolled, which include HBeAg positive and negative Chronic hepatitis B(CHB)group.

DETAILED DESCRIPTION:
Generic emtricitabine(FTC) has been approved for treatment of naive chronic hepatitis B(CHB) patients in China. Yet data are limited for this agent in children paitients. The investigators design this trial to test the effect of FTC in Chinese children CHB which including naive HBeAg positive and Negative CHB patients.

ELIGIBILITY:
Inclusion Criteria:

* Children with body weight ≥ 33 kg and who can swallow entire emtricitabine capsle(200mg)
* HBsAg positive for more than 6 months
* HBeAg positive patients: HBV DNA ≥ 5log10 copies/ml
* HBeAg positive patients: ALT≥2×ULN;or liver biopsy G≥2;or liver biopsy S ≥2;or liver biopsy Knodell HAI ≥ 4
* HBeAg negative patients: HBV DNA ≥ 4log10 copies/ml
* HBeAg positive patients: ALT≥2×ULN;or liver biopsy G≥2;or liver biopsy S ≥2;or liver biopsy Knodell HAI ≥ 4
* Nucleoside/nucleotide naive patients

Exclusion Criteria:

* - Diagnosed HCC with AFP and ultrasound, CT or MRI
* Creatine >130μmol/L or Ccr < 70mL/min
* Hemoglobin <100g/L
* Neutrophils <1.5E+9/L
* PLT<80E+9/L
* Coinfected with HAV,HEV,HCV,HDV or HIV
* ANA > 1:100
* Uncontrolled cardiovascular diseases, kidney diseases,lung diseases, neurological diseases, digestive diseases,metabolic disorders, immune-compromised diseases or cancer
* Drug abuse or alcohol addiction
* Previous history of taking agents of lamivudine, adefovir, tenofovir entecavir or telbivudine
* Long-term use of immunosuppressor or immunomodulator 6 months before enrollment to this trial
* Underwent liver transplantation or liver transplantation in schedule
* Allergic to nucleoside or nucleotide analogues
* Pregnancy or in breastfeeding

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
virological response rate | week 48
  HBV DNA < 500 copies/ml

SECONDARY OUTCOMES:
HBV DNA negativity rate | week 24
  HBV DNA < 500 copies/ml
HBV DNA decrease level | week24 and 48
  HBV DNA decrease compared with baseline（log10 copies/ml）
biochemical response | week 24 and 48
  ALT normalization
HBeAg loss | week 24 and 48
  HBeAg loss in HBeAg positive group
HBeAg seroconversion | week 24 and 48
  HBeAg seroconversion in HBeAg positive group
HBeAg reversion | week 24 and 48
  HBeAg positive in Baseline HBeAg negativie group patients
HBsAg loss | week 24 and 48
  HBsAg loss
HBsAg seroconversion | week 24 and 48
  HBsAg loss and anti-HBs positive
HBV genetic resistance to emtricitabine | week 24 and 48
  HBV genetic resistance to emtricitabine
adverse event | week 24 and 48
  type and rate of adverse events;type and rate of severe adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cheng, M.D., Principal Investigator — Asian Pacific Alliance of Liver Diseases, Beijing

REFERENCES:
- [Background] Gish RG, Leung NW, Wright TL, Trinh H, Lang W, Kessler HA, Fang L, Wang LH, Delehanty J, Rigney A, Mondou E, Snow A, Rousseau F. Dose range study of pharmacokinetics, safety, and preliminary antiviral activity of emtricitabine in adults with hepatitis B virus infection. Antimicrob Agents Chemother. 2002 Jun;46(6):1734-40. doi: 10.1128/AAC.46.6.1734-1740.2002. PMID 12019083